CLINICAL TRIAL: NCT07143370
Title: Microbial Colonization in 3D Printed Orthodontic Clear Aligners
Brief Title: Microbial Colonization in Three Dimensional (3D) Printed Orthodontic Clear Aligners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Aron Aliaga del Castillo, Clinical Assistant Professor of Dentistry, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00268846
Record Dates: First submitted 2025-08-07; First posted 2025-08-27 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Orthodontic Aligner; Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- 3D printed clear aligner TC-85 (Experimental): Results compiled for this aligner from all orders of aligner assignments.
  Interventions: Device: Thermoformed clear aligner; Device: 3D printed clear aligner TC-85; Device: 3D printed clear aligner TA-28
- 3D printed clear aligner TA-28 (Experimental): Results compiled for this aligner from all orders of aligner assignments.
  Interventions: Device: Thermoformed clear aligner; Device: 3D printed clear aligner TC-85; Device: 3D printed clear aligner TA-28
- Thermoformed clear aligner (Experimental): Results compiled for this aligner from all orders of aligner assignments.
  Interventions: Device: Thermoformed clear aligner; Device: 3D printed clear aligner TC-85; Device: 3D printed clear aligner TA-28

INTERVENTIONS:
Device: Thermoformed clear aligner — All participants will receive a thermoformed aligner fabricated from polyethylene terephthalate glycol (PETG) material. This aligner is made from using an intraoral scan to print a 3D model of their maxillary dentition, that is then used for the thermoforming process. This aligner will be worn 20-22 hrs/day for 1 week.
Device: 3D printed clear aligner TC-85 — All participants will receive a 3D printed aligner fabricated from TC-85 resin. This aligner will be made using an Stereolithography (STL) file from their intraoral scan to design the clear aligner and then will be fabricated using the SprintRay Pro 95 S printer. This aligner will be worn 20-22 hrs/day for 1 week.
Device: 3D printed clear aligner TA-28 — All participants will receive a 3D printed aligner fabricated from TA-28 resin. This aligner will be made using an STL file from their intraoral scan to design the clear aligner and then will be fabricated using the SprintRay Pro 95 S printer. This aligner will be worn 20-22 hrs/day for 1 week.

SUMMARY:
This study is being done to compare conventional clear aligners with 3D printed clear aligners to assess if there is any significant difference between the microbial colonization of these appliances. The 3D printed aligner material and conventional aligner materials are being used for investigational purposes and have been approved for their use in fabricating clear aligners for orthodontic tooth movement, but not for the purposes of our study, which is for the fabrication of clear passive aligners to assess microbial colonization.

ELIGIBILITY:
Inclusion Criteria:

* Participants are in the permanent dentition
* Participants can understand written English instructions
* Participants have no history of smoking
* Participants will not undergo any active orthodontic treatment.

Exclusion Criteria:

* Periodontal disease/gingivitis or craniofacial anomalies.
* Severe tooth crowding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-09-02 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Microbial colonization of the tooth surface | 1 week Immediately following aligner wear
  Assessed using a swab to the tooth surface (three times, once for each aligner)
Microbial composition of inner surface biofilm of aligners | 1 week Immediately following aligner wear
  Assessed using a swab of the inside of each aligner (three times, once for each aligner)

SECONDARY OUTCOMES:
Patient perception of clear aligners | Approximately 6 weeks
  Assessed using a 11 question survey (9 questions use a likert like scale of 0(poor)-10(excellent))

CONTACTS AND LOCATIONS:
Overall Officials: Aron Aliaga del Castillo, DDS, MS, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No